CLINICAL TRIAL: NCT03947619
Title: Primary Unloading and Delayed Reperfusion in ST-Elevation Myocardial Infarction: The STEMI-DTU Trial
Acronym: DTU-STEMI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abiomed Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: The STEMI-DTU Trial
Record Dates: First submitted 2019-05-06; First posted 2019-05-13 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: ST Elevation (STEMI) Myocardial Infarction of Anterior Wall
Keywords: Anterior STEMI; ST-Elevated MI; Cardiac Unloading
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: A prospective, multicenter, randomized, controlled open-label two-arm trial with an adaptive design
Who Masked: Outcomes Assessor
Masking Description: Blinding of the operator and patient is not possible given the nature of the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Experimental (Experimental): Subjects randomized to the experimental arm will have their heart unloaded for 30 minutes on the Impella CP® device prior to PCI.
  Each site is required to have one "roll-in" per arm to test the study protocol before beginning enrollment.
  Interventions: Device: Impella CP® placement prior to reperfusion with Primary PCI
- Control (No Intervention): Primary PCI. Each site is required to have one "roll-in" per arm to test the study protocol before beginning enrollment.

INTERVENTIONS:
Device: Impella CP® placement prior to reperfusion with Primary PCI — Subjects randomized to the experimental arm, will undergo Impella CP® placement through a femoral arterial sheath and the Impella device will be activated to unload the left ventricle.
  Arms: Experimental

SUMMARY:
The purpose of this research study is to evaluate whether using the the IMPELLA® CP System temporary circulatory assist device for 30 minutes prior to a catheterization procedure has the potential to reduce the damage to the heart caused by a heart attack, compared to the current standard of care.

DETAILED DESCRIPTION:
To demonstrate the safety and effectiveness of primary Left Ventricular unloading and a thirty-minutes delay to reperfusion vs. current standard of care in reducing infarct size and heart failure-related clinical events in patients presenting with anterior ST-Elevation Myocardial Infarction.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85 years
2. First myocardial infarction
3. Acute anterior STEMI with ≥2 mm in 2 or more contiguous anterior leads or ≥ 4 mm total ST segment deviation sum in the anterior leads V1-V4 AND anterior wall motion abnormality noted on a diagnostic quality left ventriculogram or echocardiogram
4. Patient presents to the enrolling hospital where the index procedure will be performed between 1 - 6 hours after onset of continuous ischemic pain
5. Patient indicated for Primary PCI
6. Patient or the patient's Legally Authorized Representative (where applicable) has signed Informed Consent

Exclusion Criteria:

1. Patient transferred from an outside hospital where invasive coronary procedure was attempted (including diagnostic catheterization)
2. Unwitnessed cardiac arrest OR ≥30 minutes of CPR prior to enrollment OR any cardiac arrest with impairment in mental status, cognition, or any global or focal neurological deficit
3. Administration of fibrinolytic therapy within 24 hours prior to enrollment
4. Cardiogenic shock defined as: systemic hypotension (systolic BP <90 mmHg or the need for inotropes/pressors to maintain a systolic BP >90mmHg) plus one of the following: any requirement for pressors/inotropes prior to arrival at the catheterization laboratory, clinical evidence of end organ hypoperfusion or use of IABP or any other circulatory support device
5. Inferior STEMI or suspected right ventricular failure
6. Any contraindication or inability to place the Impella, including peripheral vascular disease, tortuous vascular anatomy, femoral bruits or absent pedal pulses
7. Severe aortic stenosis
8. Acute cardiac mechanical complication: LV free wall rupture OR Interventricular septum rupture OR Acute mitral regurgitation
9. Suspected or known pregnancy
10. Suspected systemic active infection
11. History or known hepatic insufficiency prior to catheterization
12. On renal replacement therapy
13. COPD with home oxygen therapy or on chronic steroid therapy
14. Known or evidence of prior myocardial infarction, including pathologic Q waves in non-anterior leads
15. Prior CABG or LAD PCI
16. History of heart failure (documented history of EF <40% or documented hospitalization for HF within one (1) year prior to screening)
17. Prior aortic valve surgery or TAVR
18. Left bundle branch block (new or old)
19. History of stroke/TIA within the prior 3 months, any history of Intracranial Hemorrhage or any permanent neurological deficit
20. History of bleeding diathesis or known coagulopathy (including heparin-induced thrombocytopenia), any recent GU or GI bleed, or will refuse blood transfusions
21. Patient on systemic anticoagulation pre-procedure (including factor Xa inhibitors, thrombin inhibitors, warfarin)

    Known contraindication to:
22. Undergoing MRI or use of gadolinium, [CrCl<30 ml/min, non-compatible implant, claustrophobia]
23. Heparin, pork, pork products or contrast media
24. Receiving a drug-eluting stent
25. Participation in the active treatment or follow-up phase of another clinical study of an investigational drug or device which has not reached its primary endpoint.
26. Any organ condition, concomitant disease (e.g., psychiatric illness, severe alcoholism, or drug abuse, severe cancer, hepatic or kidney disease), with life expectancy of ≤2 years or other abnormality that itself, or the treatment of which, could interfere with the conduct of the study or that, in the opinion of the Investigator and/or Sponsor's medical monitor, would pose an unacceptable risk to the patient in the study.
27. Subject has other medical, social, or psychological problems that, in the opinion of the Investigator, compromises the subject's ability to give written informed consent and/or to comply with study procedures, including follow-up CMRs.
28. Subject belongs to a vulnerable population [Vulnerable patient populations are defined as Individuals with mental disability, persons in nursing homes, children, impoverished persons, homeless persons, nomads, refugees, prisoners, and those permanently incapable of giving informed consent. Vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the Sponsor, and members of the armed forces.

    * A pregnancy test will be conducted prior to enrollment if required by Institutional Review Board (IRB), Regional Ethics Board (REB), local Ethics Committee (EC) or competent authority.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 527 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Infarct Size | 3-5 days post-procedure
  Infarct size normalized to the left ventricular mass, evaluated using Cardiac Magnetic Resonance (CMR) imaging

SECONDARY OUTCOMES:
Infarct Size, as a percent of Left Ventricular Mass | 3-5 days
  Efficacy- Composite clinical secondary endpoint, Compared between groups in a hierarchical order using the Finkelstein-Schoenfeld statistic.
Impella CP® related Major Bleeding and Major Vascular complications | 30 Days
  Efficacy (Cardiogenic Shock)- Composite clinical secondary endpoint. Compared between groups in a hierarchical order using the Finkelstein-Schoenfeld statistic. Secondary Safety (Major Bleeding and Vascular Complications); with pre-specified performance goals.
Cardiogenic Shock, CV mortality, Heart Failure, LVAD or Heart Transplant and ICD or CRT Placement | 12 Months
  Efficacy- Composite clinical secondary endpoint. Compared between groups in a hierarchical order using the Finkelstein-Schoenfeld statistic.

CONTACTS AND LOCATIONS:
Overall Officials: William O'Neill, MD, Principal Investigator — Henry Ford Hospital; Norman Mangner, Prof. Dr. med. habil., Principal Investigator — Heart Center Dresden
Locations (63):
- United States (46):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - HonorHealth Research Institute, Scottsdale, Arizona
  - The University of Arizona, Tucson, Arizona
  - Emanate Health Intercommunity Hospital / Valley Clinical Trials, Inc., Covina, California
  - Riverside Community Hospital, Riverside, California
  - St. Anthony Hospital, Lakewood, Colorado
  - Hartford Health Care, Hartford, Connecticut
  - Christiana Care Health Services, Newark, Delaware
  - George Washington University, Washington D.C., District of Columbia
  - BayCare Cardiology - Morton Plant Hospital, Clearwater, Florida
  - Baptist Health Research Institute, Jacksonville, Florida
  - Tallahasse Research Institute, Tallahassee, Florida
  - AdventHealth - Tampa, Tampa, Florida
  - Northside Hospital, Atlanta, Georgia
  - Wellstar/Kennestone Hospital, Marietta, Georgia
  - North Shore University Health System, Evanston, Illinois
  - Midwest Cardiovascular Institute, Naperville, Illinois
  - OSF Saint Francis, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Mercy Iowa Heart, West Des Moines, Iowa
  - Tufts Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension St. John Hospital, Detroit, Michigan
  - Spectrum, Grand Rapids, Michigan
  - Hackensack Medical Center, Hackensack, New Jersey
  - Hackensack Meridian Mountainside Medical Center, Montclair, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - Presbyterian Heart Research Group, Albuquerque, New Mexico
  - University of Buffalo Hospital, Buffalo, New York
  - Northwell Health, Manhasset, New York
  - NYU School of Medicine, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Prisma Health, Columbia, South Carolina
  - Greenville Health System, Greenville, South Carolina
  - Ballad Health - Wellmont CVA Institute, Kingsport, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Centennial Medical Center, Nashville, Tennessee
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Methodist Hospital, San Antonio, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - West Virginia University Hospital, Morgantown, West Virginia
- Canada (3):
  - University of Calgary, Calgary, Alberta
  - Hamilton Health Science, Hamilton, Ontario
  - University of Ottawa Heart Institue, Ottawa, Ontario
- Germany (8):
  - University Hospital Würzburg, Würzburg, Bavaria
  - University Hospital Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - West German Heart Center Essen, Essen, North Rhine-Westphalia
  - Krankenhaus der Barmherzigen Brüder Trier, Trier, Rhineland-Palatinate
  - Heart Center Dresden, Dresden, Saxony
  - Universitätsklinikum Jena, Jena
  - University Hospital of Marburg, Marburg
  - Heinrich-Braun-Klinikum Zwickau, Zwickau
- Italy (4):
  - Ospedale Policlinico San Martino, Genoa, Liguria
  - San Raffaele, Milan, Lombardy
  - Azienda Ospedaliera Universitaria Integrata Di Verona, Verona, Veneto
  - Humanitas Clinical & Research Hospital, Rozzano
- Luzerner Kantonsspital, Lucerne, Switzerland
- Harefield Hospital, Harefield, United Kingdom